CLINICAL TRIAL: NCT01326390
Title: Impact of C-arm CT in Patients With Decreased Renal Function Undergoing Transhepatic Arterial Chemoembolization (TACE) for the Treatment of Hepato-Cellular Carcinoma
Brief Title: Impact of C-arm CT in Decreased Renal Function Undergoing TACE for Tx of Hepato-Cellular Carcinoma
Status: Terminated | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: HEP0035; SU-07012010-6469 (Other: Stanford University)
Record Dates: First submitted 2010-07-06; First posted 2011-03-30 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Kidney (Renal Cell) Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Cerebral Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: dTA/dBA C-arm fluoroscopy system with Dyna CT — C-arm CT of the liver; state-of-the-art flat panel detector on a ceiling or floor mounted C-arm gantry
  Other Names: X-ray image intensifier; Siemens Angiography systems
Procedure: DSA arteriogram- hepatic arteries — Standard of care
  Other Names: Angiography; arteriography
Procedure: CO2 aortogram — Standard of care
  Other Names: Aortography

SUMMARY:
Impact on contrast dose or total volume of contrast required to effectively treat the targeted tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be affected by HCC
2. Patients must have diminished renal function (GFR<60 ml/min/1.73m^2)
3. Patients must be 18 years old or older
4. Patients must have received an abdominal CT, PET/CT scan or MRI, completed prior to the TACE procedure.
5. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Subjects under the age of 18
2. Patients currently on dialysis
3. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients we are seeking will already have been scheduled to undergo liver Transhepatic arterial chemoembolizationWorld Health Organization treatment using C-arm CT as the imaging guidance (with limited Digital Subtraction angiography as needed).
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2010-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients that develop renal failure (defined as a decline of renal function, as measured by glomerular filtration rate, of 25% or more from pre-procedural) | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nishita N. Kothary, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States